CLINICAL TRIAL: NCT02291068
Title: Psychological Flexibility and Effectiveness of Psychotherapy Treatment in Patients With Adjustment Disorder
Brief Title: Psychological Flexibility and Effectiveness of Psychotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TelAvivSMO
Record Dates: First submitted 2014-10-20; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Adjustment Disorder
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- psychotherapy treatment (Other): 3 months long (12 sessions) dynamic psychotherapy.
  Interventions: Behavioral: psychotherapy treatment

INTERVENTIONS:
Behavioral: psychotherapy treatment — 3 months long (12 sessions) dynamic psychotherapy. The dynamic psychotherapeutic technique which will be applied in the current research is derived from Malan's focused, brief psychodynamic psychotherapy (Malan 1976) and from the literature specifying psychodynamic psychotherapies distinctive techniques (Shedler 2010). The principle of this treatment is a time limited intervention in which the primary objective is to enhance the patient's insights regarding repetitive conflicts. As psychodynamic psychotherapy is suitable for all kinds of adjustment disorders, no special adjustment in the course of therapy was made for the different subtypes (Cabaniss et al. 2011).

SUMMARY:
The Objectives of the current research is to evaluate whether psychological flexibility influences psychotherapy outcomes in patients with adjustment disorder and depression. If indeed this is the case, we would be able to identify risk factors for low adjustment- such as low psychological flexibility, and develop psychotherapy that would try to enhance this ability.

DETAILED DESCRIPTION:
Subjects will be recruited from the Psychiatric daycare center at the Tel-Aviv Souraski Medical Center, serving the broader Tel-Aviv municipal area. Referrals to the department will be screened for eligibility to participate in the study according to the study's inclusion and exclusion criteria. Inclusion criteria would be adjustment disorder as the referral cause, age ranging from 20 to 65 years old and Hebrew speaking. Patients with major depression, a psychotic disorder, alcohol or drug dependence will be excluded. All participants will sign a written informed consent. The diagnosis of adjustment disorder will be conﬁrmed by an open clinical interview followed by a Structured Clinical Interview for DSM-IV SCID-IV (Shalev et al. 1994; First et al. 1995).

Before starting the psychotherapy treatment, the patients will fill a psychological flexibility questionnaire (PFQ) and well-being questionnaire (MHI), in order to evaluate their psychological flexibility and well-being baseline. At the end of the psychotherapy treatment, they will fill the questionnaires again. Also, their therapists will evaluate the patients' levels of adjustment disorder or depression before and after the therapy.

ELIGIBILITY:
Inclusion Criteria:

Adjustment disorder as the referral cause, age ranging from 20 to 65 years old and Hebrew speaking. The diagnosis of adjustment disorder will be conﬁrmed by an open clinical interview followed by a Structured Clinical Interview for DSM-IV SCID-IV (Shalev et al. 1994; First et al. 1995).

Exclusion Criteria:

Patients with major depression, a psychotic disorder, alcohol or drug dependence will be excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of psychotherapy treatment will be measured by the SCID-IV, CGS and CGI measures by the therapists | end of the psychotherapy treatment- an expected average of 3 months after starting therapy
  Psychotherapy outcomes will be evaluated by the patients and therapists, using a number of measures. First, the therapists would use the SCID-IV, as they did at the beginning of the treatment. Second, they would fill out a CGS and CGI questionnaires.

SECONDARY OUTCOMES:
Well being will be measured by the Mental Health Inventory (MHI: Veit and Ware 1983) | Baseline and at the end of the psychotherapy treatment-an expected average of 3 months after starting therapy
  The Mental Health Inventory (MHI: Veit and Ware 1983), a self-report questionnaire which measures psychological distress and well-being, psychiatric symptoms, and clinician rating of illness severity, will be used to measure psychological distress and well-being in the past month.
Therapeutic Alliance will be measured by the The Working Alliance Inventory-Short Revised (WAI-SR) (Munder et al., 2010) | end of the psychotherapy treatment- an expected average of 3 months after starting therapy
  The Working Alliance Inventory-Short Revised (WAI-SR) (Munder, Wilmers, Leonhart, Linster, & Barth, 2010) is a measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. It is a self-report questionnaire, which includes 12 items on 1-5 scale. A high score indicates a better therapeutic alliance. The questionnaire was translated to Hebrew and back-translated by the researchers of the current research.
Psychological Flexibility will be measured by the Psychological Flexibility Questionnaire (PFQ) (Ben-Itzhak et al., 2014). | Baseline and at the end of the psychotherapy treatment-an expected average of 3 months after starting therapy
  Psychological Flexibility Questionnaire (PFQ) (Ben-Itzhak, Bluvstein, & Maor, 2014), which includes 20 items 20, divided to 5 factors, each relating to a significant domain of psychological flexibility: (1) positive perception of change; (2) characterization of the self as flexible; (3) self-characterization as open and innovative; (4) a perception of reality as dynamic and changing, and (5), a perception of reality as multifaceted.

CONTACTS AND LOCATIONS:
Overall Officials: Shulamit Ben Itzhak, Dr, Principal Investigator — shulamitb@tlvmc.gov.il